CLINICAL TRIAL: NCT01728194
Title: White Matter and Emotional and Cognitive Control in Late-Onset Depression
Brief Title: Emotional and Cognitive Control in Late-Onset Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1205012392; 1R01MH097735-01 (NIH)
Record Dates: First submitted 2012-11-12; First posted 2012-11-16 (Estimated); Results first posted 2020-10-06 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-09

CONDITIONS: Depression
Keywords: Depression; Depressive Disorder; Behavioral Symptoms; Mood Disorders; Mental Disorders; Escitalopram; Central Nervous System Agents; Therapeutic Uses; Pharmacologic Actions; Physiological Effects of Drugs; Muscarinic Antagonists; Antidepressive Agents; Psychotropic Drugs; Serotonin Uptake Inhibitors; Neurotransmitter Uptake Inhibitors; Serotonin Agents; Magnetic Resonance Imaging, Functional; fMRI; Magnetic Resonance Imaging
MeSH Terms: conditions — Depression; Depressive Disorder; Behavioral Symptoms; Mood Disorders; Mental Disorders | interventions — Escitalopram; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Escitalopram (Experimental): Target dose 20mg for 12 weeks
  Interventions: Drug: Escitalopram; Other: Magnetic Resonance Imaging
- Control (Other): Non-psychiatric comparison participants.
  Interventions: Other: Magnetic Resonance Imaging

INTERVENTIONS:
Drug: Escitalopram — 20 mg target dose for 12 weeks
  Other Names: Lexapro; 76184942
  Arms: Escitalopram
Other: Magnetic Resonance Imaging — Structural and functional MRI of the brain for research purposes.
  Other Names: MRI

SUMMARY:
This study may help identify how abnormalities in brain systems that control the ability to ignore irrelevant information may contribute to the development of depression in older adults.

DETAILED DESCRIPTION:
Approximately half of those who develop depression in late life never had depression before. The classic view is that changes taking place in our brains as we age contribute to the development of late-onset depression. This view is supported by the relative absence of family history for those with late onset depression. This research study will recruit 70 older adults with late life depression and 70 older adults without depression. All participants will receive a sub-clinical, non-contrast (magnetic resonance imaging (MRI) scan at the beginning of the study and then again 12 weeks later at the completion of the study. The depressed older participants will also receive a Food and Drug Administration (FDA)-approved antidepressant, escitalopram (Lexapro), as treatment for their depressive symptoms over 12 weeks. This MRI study may help the researchers identify how abnormalities in brain systems that control our ability to ignore distractions, control our emotions, and anticipate reward may contribute to the development of depression in older adults. The investigators hope that the findings promote the development of tests that may improve the detection of older adults at risk for poor treatment outcomes and eventually guide the development of novel treatments for depression.

ELIGIBILITY:
Inclusion Criteria:

* Age: 60-85 years, right-handed;
* Diagnosis: Major depression, unipolar (by Structured Clinical Interview for Diagnostic and Statistical Manual (DSM)IV (SCID-R) and DSM-IV criteria);
* Age of onset of first episode ≥ 50 years with up to three depressive episodes;
* Severity of depression: A 24-Item Hamilton Depression Rating Scale (HDRS) ≥ 20.

Exclusion Criteria:

* Psychotic depression by DSM-IV, i.e., presence of delusions with a SCID-R score higher than 2;
* High suicide risk, i.e. intent or plan to attempt suicide in near future;
* Presence of any Axis I psychiatric disorder (other than unipolar major depression) or substance abuse;
* History of psychiatric disorders other than unipolar major depression or generalized anxiety disorder (bipolar disorder, hypomania, and dysthymia are exclusion criteria);
* Dementia: Diagnosis of dementia by DSM-IV;
* Mild Cognitive Impairment (MCI);
* Acute or severe medical illness, i.e., delirium, metastatic cancer, decompensated cardiac, liver or kidney failure, major surgery, stroke or myocardial infarction during the three months prior to entry; or use of drugs known to cause depression, e.g., reserpine, alpha-methyl-dopa, steroids, sympathomimetics withdrawal;
* Neurological brain disease and/or history of electroconvulsive therapy;
* History of any use of citalopram or escitalopram during the current episode or need for drugs that may interact with these agents, i.e. drug metabolized by the 2D6 P450 isoenzyme system;
* Current involvement in psychotherapy;
* Contraindications to MRI scanning including cardiac pacemaker, metallic objects and metallic implants contraindicating MRI, cardiac stent, claustrophobia;
* Inability to speak English;
* Corrected visual acuity < 20/70; Color blindness.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Faith Gunning, Ph.D., Principal Investigator — Weill Medical College of Cornell University
Locations (2):
- United States (2):
  - Weill Cornell Medical College, New York, New York
  - Weill Cornell Medical College - Westchester Division, White Plains, New York

REFERENCES:
- [Background] Victoria LW, Alexopoulos GS, Ilieva I, Stein AT, Hoptman MJ, Chowdhury N, Respino M, Morimoto SS, Kanellopoulos D, Avari JN, Gunning FM. White matter abnormalities predict residual negative self-referential thinking following treatment of late-life depression with escitalopram: A preliminary study. J Affect Disord. 2019 Jan 15;243:62-69. doi: 10.1016/j.jad.2018.09.013. Epub 2018 Sep 11. PMID 30236759
- [Derived] Oberlin LE, Victoria LW, Ilieva I, Dunlop K, Hoptman MJ, Avari J, Alexopoulos GS, Gunning FM. Comparison of Functional and Structural Neural Network Features in Older Adults With Depression With vs Without Apathy and Association With Response to Escitalopram: Secondary Analysis of a Nonrandomized Clinical Trial. JAMA Netw Open. 2022 Jul 1;5(7):e2224142. doi: 10.1001/jamanetworkopen.2022.24142. PMID 35895056
- [Derived] Respino M, Hoptman MJ, Victoria LW, Alexopoulos GS, Solomonov N, Stein AT, Coluccio M, Morimoto SS, Blau CJ, Abreu L, Burdick KE, Liston C, Gunning FM. Cognitive Control Network Homogeneity and Executive Functions in Late-Life Depression. Biol Psychiatry Cogn Neurosci Neuroimaging. 2020 Feb;5(2):213-221. doi: 10.1016/j.bpsc.2019.10.013. Epub 2019 Nov 7. PMID 31901436
- [Derived] Respino M, Jaywant A, Kuceyeski A, Victoria LW, Hoptman MJ, Scult MA, Sankin L, Pimontel M, Liston C, Belvederi Murri M, Alexopoulos GS, Gunning FM. The impact of white matter hyperintensities on the structural connectome in late-life depression: Relationship to executive functions. Neuroimage Clin. 2019;23:101852. doi: 10.1016/j.nicl.2019.101852. Epub 2019 May 3. PMID 31077981

RESULTS

PARTICIPANT FLOW:
Groups:
- MDD (Escitalopram Tx): Target dose 20mg for 12 weeks
  Escitalopram: 20 mg target dose for 12 weeks
- Control: No treatment (healthy comparison participants with no history or presence of psychiatric disorder)
Period: Overall Study
Arm/Group | MDD (Escitalopram Tx) | Control
Started | 54 | 67
Completed | 34 | 61
Not Completed | 20 | 6
Not completed — Lost to Follow-up | 4 | 3
Not completed — Physician Decision | 4 | 0
Not completed — Withdrawal by Subject | 7 | 3
Not completed — Perceived Medication Side Effects | 4 | 0
Not completed — Family Member Request | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MDD (Escitalopram Tx) | Control | Total
Number analyzed (Participants) | 54 | 67 | 121
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 9 | 19
  >=65 years | 44 | 58 | 102
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.76 (6.77) | 72.36 (6.17) | 72.09 (6.43)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 33 | 39 | 72
  Male | 21 | 28 | 49
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 0 | 6
  Not Hispanic or Latino | 48 | 67 | 115
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 5 | 7
  White | 48 | 60 | 108
  More than one race | 3 | 1 | 4
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 54 | 67 | 121
Diagnostic Status [Count of Participants; unit: Participants] — Diagnostic status based on structured clinical interview (binary outcome of "depressed" (MDD group) or "not depressed" (control group) by DSM-IV / SCID criteria)
  Participants | 54 | 67 | 121

OUTCOME MEASURES:

1. Primary Outcome: Change in Depression Severity (Measured by Montgomery Asberg Depression Rating Scale)
Description: Depression severity at baseline and week 12 in participants with MDD vs. controls, measured by score on the Montgomery Asberg Depression Rating Scale (MADRS). This measure is a clinical rating of mood with a score range from 0 to 60. Higher scores indicate greater depression severity.
Time Frame: Baseline (Study Entry / Before Tx) and Week 12 (Following Tx)
Population: 4 participants in the Escitalopram group and 4 participants in the Control group do not have follow-up MADRS data and have therefore been excluded from Week 12 analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Escitalopram: Patients diagnosed with MDD receiving 12-week Escitalopram intervention
- Control: No Intervention / Non-psychiatric comparison participants
Arm/Group | Escitalopram | Control
Number analyzed (Participants) | 54 | 67
score on a scale
  Baseline Depression Severity | 25.26 (4.65) | 1.03 (1.36)
  Week 12 Depression Severity: number analyzed (Participants) | 50 | 63
  Week 12 Depression Severity | 13.78 (9.07) | 1.08 (1.43)
Statistical Analysis 1: Comparison: Escitalopram vs Control; Test type: Other; p < 0.025, Mixed Models Analysis

2. Secondary Outcome: Change in Depression Severity (Measured by Hamilton Depression Rating Scale)
Description: Depression severity at baseline and week 12 in participants with MDD vs. controls, measured by score on the Hamilton Depression Rating Scale (HAM-D). This measure is a clinical rating of mood with a score range from 0 to 76. Higher scores indicate greater depression severity.
Time Frame: Baseline (Study Entry / Before Tx) and Week 12 (Following Tx)
Population: 4 participants in the Escitalopram group and 3 participants in the Control group do not have follow-up MADRS data and have therefore been excluded from Week 12 analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Escitalopram | Control
Number analyzed (Participants) | 54 | 67
score on a scale
  Baseline Depression Severity | 23.48 (4.45) | 1.24 (1.32)
  Week 12 Depression Severity: number analyzed (Participants) | 50 | 64
  Week 12 Depression Severity | 12.44 (8.49) | 1.52 (1.69)
Statistical Analysis 1: Comparison: Escitalopram vs Control; Test type: Other; p < 0.025, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: Baseline (Study Entry) through 12 Weeks of Treatment/Participation
Arm/Group | MDD (Escitalopram Tx) | Control
All-Cause Mortality (participants affected / at risk) | 0/54 | 0/67
Serious Adverse Events (participants affected / at risk) | 0/54 | 2/67
Other Adverse Events (participants affected / at risk) | 9/54 | 3/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MDD (Escitalopram Tx) (N=54) | Control (N=67)
Acute CVA (Surgical and medical procedures) | 0 (0) | 1 (1)
Gallbladder removal (Surgical and medical procedures) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MDD (Escitalopram Tx) (N=54) | Control (N=67)
Fall (Injury, poisoning and procedural complications) | 4 (5) | 3 (3)
Skin - Hives/Itchiness (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Elevated BP (Vascular disorders) | 2 (2) | 0 (0)
Fatigue + poor appetite (Psychiatric disorders) | 1 (1) | 0 (0)
Low libido + low mood (Psychiatric disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-07-15): https://cdn.clinicaltrials.gov/large-docs/94/NCT01728194/SAP_000.pdf
  • Study Protocol (2015-03-24): https://cdn.clinicaltrials.gov/large-docs/94/NCT01728194/Prot_001.pdf